CLINICAL TRIAL: NCT00250146
Title: Multicenter Study on the Toxicity of Gluten Traces in the Treatment of Celiac Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Associazione Italiana Celiachia (AIC) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB-2000-611
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2005-04

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Gluten; Toxicity; Small bowel morphometry
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

INTERVENTIONS:
Behavioral: Gluten (behaviour)

SUMMARY:
The purpose of this study is to evaluate the toxicity of minute doses of gluten in the treatment of celiac disease, a disorder characterized by permanent intolerance to dietary gluten.

DETAILED DESCRIPTION:
Treatment of celiac disease (CD) is based on the complete avoidance of gluten-containing products in the diet. However it is not known whether tiny amounts of gluten are harmful for patients on long-term treatment. This is an important issue, as even a strict gluten-free diet (GFD) is usually contaminated by traces of gluten, e.g. in wheat starch and processed food. The aim of this study is to investigate the toxicity of the prolonged ingestion of gluten traces in treated CD patients. This is a prospective, placebo-controlled, double-blind study. Patients are adults with biopsy-proven CD on treatment with the GFD for at least 2 years. During the study period their background daily gluten intake is kept lower than 5 mg. After baseline evaluation, patients continue their GFD and are assigned to ingest 0 mg, 10 mg or 50 mg of daily gluten (incorporated in a capsule) for 90 days. The following evaluations are performed both at baseline and after the micro-challenge: clinical, serological (anti-transglutaminase and antigliadin antibodies), and small intestine histology.

ELIGIBILITY:
Inclusion Criteria:

adults with biopsy-proven celiac disease on a gluten-free diet for at least 2 years and in apparent good health -

Exclusion Criteria:

1. patients younger than 18 years old;
2. poor compliance to the gluten-free diet;
3. abnormal results at the baseline evaluation (positivity of anti-tissue transglutaminase (tTG) antibodies and/or definitely abnormal small intestinal biopsy;
4. associated conditions, such as selective IgA deficiency or other autoimmune diseases -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2001-02; Study Completion 2005-03

PRIMARY OUTCOMES:
Villous Height/Crypt Depth ratio on small intestinal biopsy
Intraepithelial lymphocyte coun on small intestinal biopsy
changes in serum IgA class anti-trasnglutaminase antibodies
changes in serum IgG class anti-gliadin antibodies
clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, M.D., Principal Investigator — Department of Pediatrics, Università Politecnica delle Marche, Ancona, Italy
Locations (1):
- University Department of Pediatrics, Ancona, Ancona, Italy